CLINICAL TRIAL: NCT01384682
Title: Randomised, Openlabel Study Evaluating Efficacy and Safety of Maraviroc as a Switch for Either NRTI or PI/r in HIV-1 Infected Individuals With Stable, Well-Controlled Plasma HIV-RNA While Taking Their First N(t)RTI + PI/r Regimen of cART
Brief Title: Maraviroc Switch Collaborative Study
Acronym: MARCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: ViiV Healthcare (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-01-MAR
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: HIV
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No change (No Intervention): continue their current cART regimen
- Replace N(t)RTI drugs with Maraviroc (Active Comparator): Replace N(t)RTI drugs with MVC at a dose of 150mg bid (MVC 300mg bid can be used at the discretion of the Investigator if the PI/r is fosamprenavir/r) and continue the PI/r
  Interventions: Drug: Maraviroc
- Replace PI/r drugs with Maraviroc (Active Comparator): Replace PI/r drugs with MVC at a dose of 300mg bid and continue 2N(t)RTI.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc is a marketed drug for the treatment of HIV-infection. Maraviroc will be supplied in two different oral dose forms, 150mg and 300mg given twice a day. The drug will be dosed according to the recommendations in the product label i.e. with PI/r the dose is 150mg bid except, Maraviroc 300mg bid can be used at the discretion of the investigator if the PI/r is fosamprenavir/r; those randomised to the 2N(t)RTI arm, will receive Maraviroc 300mg bid. Patients randomised to receive Maraviroc will be provided with bottles of Maraviroc which contain a 30-day supply.
  Arms: Replace N(t)RTI drugs with Maraviroc; Replace PI/r drugs with Maraviroc

SUMMARY:
MARCH is an international, multicentre trial planning to enroll 380 HIV-1 infected patients who are currently on 2N(t)RTI + PI/r regimen and virologically suppressed. Participants will be randomized (1:2:2) to one of three treatment groups: to continue their current treatment regimen, maraviroc dose at 150 mg twice daily with PI/r, or maraviroc at 300 mg twice daily with 2N(t)RTI. As the participants population have HIV RNA <200 copies/mL, the phenotypic assessment of tropism cannot be used to determine tropism, instead we will employ the genotypic assessment of tropism by sequencing the V3 loop of the HIV envelope. The main aim of this study is to investigate whether switching to maraviroc, in combination with either RTI or PI/r, is as good at keeping the HIV viral load undetectable as the combination of RTI with PI/r. The other aim is to see if switching to these combinations with maraviroc will improve some of the side effects that can be seen when people take combination therapy including RTI and PI/r.

The study hypothesis is that in stable, virologically suppressed (plasma HIV-RNA <200 copies/mL) patients with no history of prior virological failure, a switch to either MVC dosed at 300mg twice daily (bid) combined with the same 2N(t)RTI backbone regimen or MVC dosed at 150mg twice daily (bid) with the current PI/r (or 300mg bid at the discretion of the investigator if the PI/r is fosamprenavir/r) provides similar (non-inferior) antiretroviral efficacy compared to continuation of the current 2N(t)RTI + PI/r regimen.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection by a licensed diagnostic test at any time prior to study entry
* Age >18 years
* HIV-1 RNA <200 copies/mL plasma for at least 24 weeks
* Stable (>24 weeks) ART including two N(t)RTIs and a PI/r
* No evidence of any primary HIV genotypic mutations in HIV reverse transcriptase or protease for all patients with available resistance testing results conducted prior to cART and/or during viral rebound/failure
* Provision of written, informed consent.

Exclusion Criteria:

* CXCR4 or CCR5/CXCR4 dual tropic HIV tropism or a non-reportable tropism result based on assessment using proviral DNA
* Anticipated need to modify current cART regimen for toxicity management in the next 6 months
* The following laboratory criteria,

  1. absolute neutrophil count (ANC) <750 cells/µL
  2. haemoglobin <8.0 g/dL
  3. platelet count <50,000 cells/µL
  4. serum AST, ALT >5 x upper limit of normal (ULN)
* Active hepatitis B co-infection
* Pregnant women or nursing mothers
* Current use of any prohibited medications as described in product specific information.
* Hypersensitivity to soy or peanuts
* Acute therapy for serious infection or other serious medical illness (in the judgement of the site Principal Investigator) requiring systemic treatment and/or hospitalisation
* Use of immunomodulators (e.g. systemic corticosteroids, recombinant interleukin-2, interferon) within 30 days prior to screening
* Patients with current alcohol or illicit substance use that in the opinion of the site Principal Investigator would conflict with any aspect of the conduct of the study
* Patients unlikely to be able to remain in follow-up for the protocol-defined period
* Prisoners or subjects who are compulsorily detained (involuntary incarcerated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The comparison of the switch arms to control arm of proportions of participants with HIV RNA <200 copies/mL 48 weeks after randomisation. | 48 weeks after randomization

SECONDARY OUTCOMES:
Virological endpoints: proportion of participants with plasma HIV-1 RNA<50 copies/ml | 48 weeks from randomization
  A number of secondary endpoints will be examined at or through to week 48 in this protocol. These will include, but not be limited to the following:
  Virologic; Immunologic and biomarkers; Clinical; Metabolic and body composition; Safety; Adherence; Quality of Life and Resistance endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: David A Cooper, AO, Principal Investigator — Kirby Institute, University of New South Wales
Locations (51):
- Argentina (8):
  - Fundacion IDEAA, Buenos Aires, Buenos Aires
  - Hospital Nacional Prof Alejandro Posadas, El Palomar, Buenos Aires
  - Hospital Dr Diego Paroissien, Isidro Casanova, Buenos Aires
  - FUNCEI, Buenos Aires, Buenos Aires F.D.
  - Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Hospital G de Agudos JM Ramos Mejia, Buenos Aires, Buenos Aires F.D.
  - CAICI, Rosario, Santa Fe Province
  - Hospital Privado- Centro Medico Cordoba, Córdoba
- Australia (10):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Gladstone Road Medical Centre, Bisbane, Queensland
  - Brisbane Sexual Health and HIV Service (formerly AMU), Brisbane, Queensland
  - Nambour General Hospital, Nambour, Queensland
  - O'Brien Street Practice, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
- Canada (4):
  - Southern Alberta Clinic, Calgary, Alberta
  - University Health Network/Toronto General Hospital, Toronto, Ontario
  - Canadian Immunodeficiency Research Collaborative (CIRC) lnc (Maple Leaf Clinic), Toronto, Ontario
  - Clinic Opus/Lori, Montreal, Quebec
- Fundación Arriarán, Santiago, Santiago RM, Chile
- Service Maladies infectieuses et Tropicales CHR ORLEANS La SOURCE, Orléans, France
- Germany (7):
  - Johann Wolfgang Goethe-University Hospital, Medical HIVCENTER, Frankfurt, Frankfurt Am Main
  - Gemeinschaftspraxis Jessen Jessen Stein, Berlin, State of Berlin
  - Dienstleistung centre ID (Baumgarten, MIB medical center for infectious diseases), Berlin
  - University of Bonn, Med J. Immunologische Siudienzenirale, Bonn
  - Klinikum der Universitat Zu Koln, Cologne
  - Universitätsklinikum Düsseldorf, Klinik für Gastroenterologie, Hepatologie und Infektiologie-MX- Amb, Düsseldorf
  - Klinik für Immunologie und Rheumatologie, Medzinische Hochschule Hannover, Hanover
- Mater Misericordiae University Hospital, Dublin, Dublin, Ireland
- Nagoya Medical Center, Nagoya, Japan
- Mexico (3):
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Hospital General de Leon, León
  - INCMNSZ, Mexico City
- Wojewodzki Szpital Zakazny Centrum Diagnostyki i Terapii AIDS, Warsaw, Warsaw, Poland
- Spain (8):
  - Hospital Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Clínic de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Regional Carlos Haya de Málaga, Málaga, Malaga
  - Hospital La Paz,, Madrid
  - Hospital Principe de Asturias, Madrid
  - Virgen Del Rocio University Hospital, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Chulalongkorn University Hospital, Bangkok, Bangkok, Thailand
- United Kingdom (5):
  - St. Mary's Hospital, Imperial College, London, London
  - St. Thomas's Hospital, London, London
  - Western General Hospital, Edinburgh, Lothian
  - Brighton & Sussex University NHS Trust, Brighton, Sussex
  - Coventry and Warwickshire Partnership Trust, Coventry, Warwickshire

REFERENCES:
- [Derived] Pett SL, Amin J, Horban A, Andrade-Villanueva J, Losso M, Porteiro N, Sierra Madero J, Belloso W, Tu E, Silk D, Kelleher A, Harrigan R, Clark A, Sugiura W, Wolff M, Gill J, Gatell J, Fisher M, Clarke A, Ruxrungtham K, Prazuck T, Kaiser R, Woolley I, Arnaiz JA, Cooper D, Rockstroh JK, Mallon P, Emery S; Maraviroc Switch (MARCH) Study Group. Maraviroc, as a Switch Option, in HIV-1-infected Individuals With Stable, Well-controlled HIV Replication and R5-tropic Virus on Their First Nucleoside/Nucleotide Reverse Transcriptase Inhibitor Plus Ritonavir-boosted Protease Inhibitor Regimen: Week 48 Results of the Randomized, Multicenter MARCH Study. Clin Infect Dis. 2016 Jul 1;63(1):122-32. doi: 10.1093/cid/ciw207. Epub 2016 Apr 5. PMID 27048747
- [Derived] Tu E, Swenson LC, Land S, Pett S, Emery S, Marks K, Kelleher AD, Kaye S, Kaiser R, Schuelter E, Harrigan R; MARCH Laboratory Group and the MARCH Study Group. Results of external quality assessment for proviral DNA testing of HIV tropism in the Maraviroc Switch collaborative study. J Clin Microbiol. 2013 Jul;51(7):2063-71. doi: 10.1128/JCM.00510-13. Epub 2013 Apr 17. PMID 23596247
- See also: Kirby Institute for infection and immunity in society homepage - click here for more information on the MARCH study. — http://www.kirby.unsw.edu.au